CLINICAL TRIAL: NCT03411473
Title: A Phase IIa Open-Label Trial of AGEN1884 in Combination With Pembrolizumab in Subjects With Chemotherapy Naïve, PD-L1 High, Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study of AGEN1884 With Pembrolizumab in 1L NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial will not proceed due to changes in the treatment landscape.
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-500-03
Record Dates: First submitted 2017-11-14; First posted 2018-01-26 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AGEN1884 with pembrolizumab (Experimental): AGEN1884 in combination with pembrolizumab
  Interventions: Biological: AGEN1884 in combination with pembrolizumab

INTERVENTIONS:
Biological: AGEN1884 in combination with pembrolizumab — AGEN1884 in combination with pembrolizumab in subjects with stage IV NSCLC whose tumors have high PD-L1 expression and no EGFR or ALK genomic tumor aberrations

SUMMARY:
A Phase IIa Open-Label Trial to Investigate the Safety, Tolerability, Pharmacokinetics, Biological, and Clinical Activity of AGEN1884 in Combination with Pembrolizumab in Subjects with Chemotherapy Naïve, PD-L1 high, metastatic Non-Small Cell Lung Cancer (NSCLC)

DETAILED DESCRIPTION:
This is a Phase IIa, open-label study, of AGEN1884 in combination with pembrolizumab in subjects with stage IV NSCLC whose tumors have high PD-L1 expression and no EGFR or ALK genomic tumor aberrations.

The study consists in two phases:

* Safety Run-in Phase
* Efficacy Phase

Subjects will be enrolled in a "3+3" Safety Run-in followed by enrollment completing the efficacy cohort. Two different dose levels of AGEN1884 may be tested in combination with the approved pembrolizumab treatment for this indication (until disease progression, unacceptable toxicity, or up to a maximum of 24 months). Each subject will stay on the dose level assigned at trial entry.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate.
2. Be ≥18 years of age.
3. Have a histologically or cytologically confirmed diagnosis of NSCLC, is stage IV, does not have an EGFR sensitizing (activating) mutation or ALK translocation, and has not received prior systemic chemotherapy treatment for their metastatic NSCLC.
4. Have measurable disease based on RECIST 1.1 as determined by the site.
5. Have a life expectancy of at least 3 months and a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status
6. Have adequate organ function as indicated by the following laboratory values:

   1. Adequate hematological function defined by absolute neutrophil count (ANC) > 1.5 x 109/L, platelet count > 100 x 109/L, and hemoglobin > 9 g/dL (without transfusions within 2 weeks of first dose).
   2. Adequate hepatic function based by a total bilirubin level < the institutional upper limit of normal (IULN), aspartate aminotransferase (AST) level < 1.5 x IULN, alanine aminotransferase (ALT) level < 1.5 x IULN, and alkaline phosphatase ≤ 2.5 ULN.
   3. Adequate renal function defined as Creatinine ≤ 1.5 x IULN OR calculated creatinine clearance > 60 mL/min for subjects with creatinine levels > 1.5 x IULN (If no local guideline is available, creatinine clearance should be calculated using the Cockcroft-Gault Method).
   4. Adequate coagulation defined by international normalized ratio (INR) or prothrombin time ≤ 1.5 x IULN (unless the subject is receiving anticoagulant therapy); and activated partial thromboplastin time (aPTT) ≤ 1.5 x IULN (unless the subject is receiving anticoagulant therapy)
   5. Adequate endocrine function defined by thyroid stimulating hormone (TSH) within normal limits. Note: if TSH is not within normal limits at baseline, the subject may still be eligible if T3 and free T4 are within normal limits.
7. Subject has no history of prior malignancy, with the exception of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy.
8. Have provided a formalin fixed tumor tissue sample from a biopsy of a tumor lesion either at the time of or after the diagnosis of metastatic disease has been made AND from a site not previously irradiated to assess for PD-L1 status.
9. The subject's tumor does not harbor an EGFR sensitizing (activating) mutation or ALK translocation.
10. The subject's tumor must have high PD-L1 expression (TPS ≥50%) as determined by an FDA-approved test.
11. Female subjects must have a negative serum pregnancy test at screening (within 72 hours of first dose of study medication) if of childbearing potential or be of non-child bearing potential.
12. If of childbearing potential, female subjects must be willing to use two adequate barrier methods throughout the study, starting with the screening visit through 120 days after the last dose of study therapy.
13. Male subjects with a female partner(s) of child-bearing potential must agree to use two adequate barrier methods throughout the trial starting with the screening visit through 120 days after the last dose of pembrolizumab is received. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.
14. Subject is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Has an EGFR sensitizing mutation and/or an ALK translocation.
2. Has received systemic therapy for the treatment of their stage IV NSCLC. Completion of treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of metastatic disease.
3. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks of the first dose of treatment.
4. Is receiving systemic steroid therapy < 3 days prior to the first dose of trial treatment or receiving any other form of immunosuppressive medication.
5. Is expected to require any other form of systemic or localized antineoplastic therapy while on trial (including maintenance therapy with another agent for NSCLC, radiation therapy, and/or surgical resection)
6. Has received prior systemic cytotoxic chemotherapy, biological therapy, OR major surgery within 3 weeks of the first dose of trial treatment; received thoracic radiation therapy of > 30 Gy within 6 months of the first dose of trial treatment.
7. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
8. Has central nervous system (CNS) metastases and/or carcinomatous meningitis identified either on the baseline brain imaging obtained during the screening period OR identified prior to signing the ICF.
9. Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (i.e., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has had an allogeneic tissue/solid organ transplant.
11. Has interstitial lung disease (ILD) OR has had a history of pneumonitis that has required oral or IV steroids.
12. Has received or will receive a live vaccine within 30 days prior to the first administration of study medication. Seasonal flu vaccines that do not contain a live virus are permitted
13. Has an active infection requiring intravenous systemic therapy.
14. Has known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
15. Has known active Hepatitis B, Hepatitis C or tuberculosis.
16. Has clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥II), or serious uncontrolled cardiac arrhythmia requiring medication.
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).
20. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit (Visit 1) through 120 days after the last dose of pembrolizumab or AGEN1884.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of DLTs in subjects in the Safety Run-in Phase of the trial | 21 days
  Occurrence of DLTs in subjects in the Safety Run-in Phase of the trial

SECONDARY OUTCOMES:
Frequency, severity, and duration of treatment-emergent AEs (TEAEs) | 116 weeks
  Frequency, severity, and duration of treatment-emergent AEs (TEAEs)
Frequency, severity, and duration of treatment-related AEs | 116 weeks
  Frequency, severity, and duration of treatment-related AEs
Confirmed BOR per RECIST 1.1 | 116 weeks
  Confirmed BOR per RECIST 1.1
Duration of response per RECIST 1.1 | 36 months
  Duration of response per RECIST 1.1
PFS time | 36 months
  PFS time
OS time | June 2020 ( When 14 patients have completed 2 years of treatment)
  OS time
Unconfirmed response at 12 weeks from first dose per RECIST 1.1 | Up to 24 months from 1st dose of treatment
  Unconfirmed response at 12 weeks from first dose per RECIST 1.1
Pharmacokinetic profile of AGEN1884 and pembrolizumab | At least 20 patients have completed 12 weeks from 1st dose of treatment
  Pharmacokinetic profile of AGEN1884 and pembrolizumab
Immunogenicity of AGEN1884 and pembrolizumab | All patients on study have completed 6 weeks from 1st dose of treatment
  Immunogenicity of AGEN1884 and pembrolizumab

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Agenus Inc.
Locations (5):
- Australia (4):
  - Mater Research, Brisbane
  - Scientia Clinical Research, Sydney
  - John Flynn Private Hospital, Tugun
  - Sydney Adventist, Wahroonga
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided